CLINICAL TRIAL: NCT02123446
Title: A Randomized, Open-label, Two-period, Two-treatment, Two-sequence, Crossover Study to Evaluate the Bioequivalence of Single Doses of Two Oral Preparations in Capsules With 250 mg of Cephalexin (Keflex® Made in Mexico by Eli Lilly y Compañía de México, S.A. de C.V. vs. Keflex® Made in Italy by Facta Farmaceutici S.p.A. for Eli Lilly y Compañía de México, S.A. de C.V.) in Fasting Healthy Volunteers
Brief Title: A Study of Cephalexin Capsules in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Investigacion Farmacologica y Biofarmaceutica, S.A. de C.V. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 15313; A3Q-ME-AFBP (Other: Eli Lilly and Company)
Record Dates: First submitted 2014-04-23; First posted 2014-04-25 (Estimated); Results first posted 2015-05-27 (Estimated); Last update posted 2015-07-15 (Estimated); Status verified 2015-06

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Cephalexin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cephalexin (Reference) (Experimental): Cephalexin manufactured in Mexico by Eli Lilly administered once orally in one of two study periods.
  Interventions: Drug: Cephalexin
- Cephalexin (Test) (Active Comparator): Cephalexin manufactured in Italy by Facta administered once orally in one of two study periods.
  Interventions: Drug: Cephalexin

INTERVENTIONS:
Drug: Cephalexin — Administered orally.
  Other Names: Keflex®

SUMMARY:
The purpose of this study is to compare two different preparations of an antibiotic called cephalexin in capsules to determine if they are essentially the same. The study has two periods. Participants will receive one preparation of cephalexin in each period. At least 7 hours will pass between the study periods. The study is expected to last about 2 days for each participant, not including screening or follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Participation will be voluntary.
* The body mass index of participants should be between 18-27.
* Participants should have a good health status.
* Limits of variation allowed within normal values at screening will be: blood pressure (seated) up to 139 millimeters of mercury (mm Hg), for systolic, and up to 89 mm Hg for diastolic; heart rate between 60 and 100 beats per minute, and respiratory rate between 14 and 20 breaths per minute.
* Hepatitis B and C and human immunodeficiency virus (HIV) negative.
* Drug abuse or alcohol detection test approximately 12 hours before administering the study medication.
* Serum pregnancy test (beta human chorionic gonadotropin) at screening and urine pregnancy test approximately 12 hours before administering the study medication.

Exclusion Criteria:

* Participants with any clinically significant abnormality in their vital sign constants recorded at screening.
* Sponsor´s and/or site employees.
* Abnormal 12 lead electrocardiogram (ECG) that in the opinion of the investigator places the participant at an unacceptable risk for study participation, Bazett corrected QR interval (QTcB) > 470 millisecond (msec) for women and > 450 msec for men.
* Participants with history of cardiovascular, renal, hepatic, muscular, metabolic, gastrointestinal diseases, including constipation, neurological, endocrine, hematopoietic diseases, or any type of anemia, asthma, mental disease, or other organic abnormalities.
* Participants with a creatinine clearance < 80 milliliter per minute (mL/min) based on the Cockcroft-Gault equation.
* Participants requiring any medication during the study, apart from the medication which is being studied.
* Participants with history of dyspepsia, gastritis, esophagitis, duodenal or gastric ulcer.
* Participants who have been exposed to medications known as hepatic enzyme inducers or inhibitors or who have been taking potentially toxic medications within the 30 days prior.
* Participants who have received any medication, including vitamins (with or without medical prescription) or herbal-based remedies 30 days (or 7 half-lives) prior to the beginning of the study.
* Participants who have been hospitalized for any condition within six months to the beginning of the study.
* Participants who have received investigational drugs within the 60 days prior to the study.
* Participants allergic to any medication, food, or substance.
* Participants who require therapy with nephrotoxic drugs.
* Participants who have donated 450 mL of blood or more within the 60 days prior to the beginning of the study.
* Participants with history of drug and alcohol abuse.
* Participants with special diet requirement for any cause.
* Participants with positive to pregnancy test or are breastfeeding.
* Participants on hormonal treatment by any route.
* Participants who have not been recorded in the page of the Comisión Federal para la Protección contra Riesgos Sanitarios (COFEPRIS).

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2014-04; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mexico City, Mexico

RESULTS

PARTICIPANT FLOW:
Groups:
- Cephalexin Dosing Sequence AB: Each participant was administered Cephalexin A formulation (Treatment A, Reference - 1 occasion) and Cephalexin B formulation (Treatment B, Test - 1 occasion).There was an interval of 1 day between doses.
- Cephalexin Dosing Sequence BA: Each participant was administered Cephalexin B formulation (Treatment B, Test - 1 occasion) and Cephalexin A formulation (Treatment A, Reference - 1 occasion).There was an interval of 1 day between doses.
Period: Period 1 (7 Days)
Arm/Group | Cephalexin Dosing Sequence AB | Cephalexin Dosing Sequence BA
Started | 14 | 14
Completed | 14 | 14
Not Completed | 0 | 0
Period: Washout Period (1 Day)
Arm/Group | Cephalexin Dosing Sequence AB | Cephalexin Dosing Sequence BA
Started | 14 | 14
Completed | 13 | 14
Not Completed | 1 | 0
Not completed — Physician Decision | 1 | 0
Period: Period 2 (7 Days)
Arm/Group | Cephalexin Dosing Sequence AB | Cephalexin Dosing Sequence BA
Started | 13 | 14
Completed | 13 | 14
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Overall Study: Each participant was administered Cephalexin A formulation (Treatment A, Reference - 1 occasion) and Cephalexin B formulation (Treatment B, Test - 1 occasion).
Arm/Group | Overall Study
Number analyzed (Participants) | 28
Age, Continuous [Mean (Standard Deviation); unit: Years] | 30.4 (8.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 28
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Mexico | 28

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics: Area Under the Concentration Versus Time Curve of Cephalexin From Time Zero to Infinity [AUC(0-∞)] of Cephalexin Following a Single Dose
Time Frame: Pre-dose, 0.25, 0.5, 0.75, 1.0, 1.25, 1.5, 1.75, 2.0, 2.5, 3.0, 3.5, 4.0, 5.0, 6.0, and 7.0 hours in each period
Population: All participants who had at least one study treatment and had evaluable pharmacokinetic (PK) data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour*microgram per milliliter(h*µg/mL)
Groups:
- Cephalexin (Reference): Cephalexin(Treatment A) manufactured in Mexico by Eli Lilly administered once orally in one of two study periods.
- Cephalexin (Test): Cephalexin(Treatment B) manufactured in Italy by Facta administered once orally in one of two study periods.
Arm/Group | Cephalexin (Reference) | Cephalexin (Test)
Number analyzed (Participants) | 25 | 25
Hour*microgram per milliliter(h*µg/mL) | 19.102 (16.751) | 19.207 (17.551)

2. Secondary Outcome: Pharmacokinetics: Maximum Concentration (Cmax) of Cephalexin
Time Frame: Pre-dose, 0.25, 0.5, 0.75, 1.0, 1.25, 1.5, 1.75, 2.0, 2.5, 3.0, 3.5, 4.0, 5.0, 6.0, and 7.0 hours in each period
Population: All participants who had at least one study treatment and had evaluable pharmacokinetic (PK) data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Microgram per milliliter(µg/ml)
Arm/Group | Cephalexin (Reference) | Cephalexin (Test)
Number analyzed (Participants) | 25 | 25
Microgram per milliliter(µg/ml) | 10.976 (24.981) | 9.710 (39.223)

3. Secondary Outcome: Pharmacokinetics: Time to Reach Maximum Observed Concentration (Tmax) of Cephalexin Following a Single Dose Maximum
Time Frame: Pre-dose, 0.25, 0.5, 0.75, 1.0, 1.25, 1.5, 1.75, 2.0, 2.5, 3.0, 3.5, 4.0, 5.0, 6.0, and 7.0 hours in each period
Population: All participants who had at least one study treatment and had evaluable PK data.
Measure: Median (Standard Deviation); unit: hours
Arm/Group | Cephalexin (Reference) | Cephalexin (Test)
Number analyzed (Participants) | 25 | 25
hours | 1.000 (0.765) | 1.000 (0.876)

ADVERSE EVENTS:
Arm/Group | Cephalexin (Reference) | Cephalexin (Test)
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/28
Other Adverse Events (participants affected / at risk) | 0/28 | 0/28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days